CLINICAL TRIAL: NCT01778621
Title: Acupuncture Treatment Versus Non-acupuncture During IVF
Brief Title: Effect of Acupuncture on Anti Mullerian Hormone and Assisted Reproduction Outcome in PCOS Patients Undergoing IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amina Altutunji (Other)
Collaborators: Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor-Investigator, Amina Altutunji, Doctor /assissted reproduction center/Union Hospital, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MINA-1978
Record Dates: First submitted 2013-01-23; First posted 2013-01-29 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: PCOS
Keywords: Acupuncture; AMH; PCOS

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Hwato®) (Experimental): 30-40 minutes acupuncture at certain acupoints that chosen according to traditional Chinese medicine and included LIV3,SP6,SP8,ST36,SP10,ST29,LI14,Ren 04;starting at follicular phase of the cycle till 2 days before oocyte picked up.
  Interventions: Device: Acupuncture(Hwato®)
- No acupuncture (No Intervention): No intervention was done for this group of patients.

INTERVENTIONS:
Device: Acupuncture(Hwato®) — acupuncture using 4cm long disposable stainless steel hair-thin needles manufactured by Suzhou medical appliance factory (China).
  Arms: Acupuncture (Hwato®)

SUMMARY:
Acupuncture at follicular phase of the cycle may improve the pregnancy rate. This study aims to compare assisted reproduction outcome between two groups of PCOS patients underwent IVF, one group received acupuncture and other group without acupuncture.

DETAILED DESCRIPTION:
Follicular phase acupuncture applied for PCOS patients underwent IVF to evaluate the effect of acupuncture on anti-mullerian hormone (AMH) and the effect on assisted reproduction outcome. It applied at certain acupoints according to the principles of traditional Chinese medicine.

ELIGIBILITY:
Inclusion Criteria::

* PCOS patients with patent one or two fallopian tubes, normal uterine cavity and partners with normal semen parameters.
* infertility
* 20-40 years
* IVF treatment -

Exclusion Criteria:

* patients with disorders that have the similar clinical presentation
* closed both tubes
* abnormal semen parameters
* intracytoplasmic sperm injection (ICSI)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate. | 13 months
  Increase in pregnancy rate

SECONDARY OUTCOMES:
Ongoing pregnancy rate | 15 months
  Increase in ongoing pregnancy rate

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gao, Ph.D., M.D., Study Director — Assisted Reproduction Center, Union Hospital
Locations (1):
- Assisted Reproduction Center, Department of Obstetrics and Gynecology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No